CLINICAL TRIAL: NCT00016692
Title: A Phase 1b Multicenter Double-Blind, Placebo-Controlled, Randomized Study on the Safety and Tolerability of Z-100 in Early HIV-1 Infected Patients
Brief Title: Safety and Tolerability of Z-100 in Patients With Early HIV Infection
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Zeria Pharmaceutical (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: B014; Zeria Protocol 85D10104
Record Dates: First submitted 2001-05-24; First posted 2001-08-31 (Estimated); Last update posted 2006-04-27 (Estimated); Status verified 2001-04

CONDITIONS: HIV Infections
Keywords: Drug tolerance; Acute Infection
MeSH Terms: conditions — HIV Infections | interventions — specific substance maruyama

INTERVENTIONS:
Drug: Z-100

SUMMARY:
The purpose of the study is to see if Z-100 (an investigational drug) treatment is safe in HIV patients who have never received treatment for their HIV, who have not been taking highly active antiretroviral therapy (HAART) for at least 8 weeks, or who have been stable on their current first or second HAART regimen for at least 12 weeks.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are HIV positive but do not show symptoms.
* Are male or female, 18 years or older.
* Have not received treatment for HIV.
* Have received treatment but have discontinued HAART for at least 8 weeks prior to screening, have had stable viral loads on at least 2 separate time points at least 1 month apart including screening, and have had stable CD4 levels on at least 2 separate time points at least 1 month apart including screening.
* Use birth control while on the study and during the follow-up period.
* Have viral loads of 2,000 to 55,000 copies/ml within 2 weeks of randomization.
* Have CD4 counts of greater than 350 cells/mm within 2 weeks of randomization.
* Have a negative serum pregnancy test within 2 weeks of randomization (women able to have children).

Exclusion Criteria

Patients will not be eligible for this study if they:

* Have failed HAART treatment.
* Have opportunistic infection or cancer.
* Have a history of tuberculosis.
* Have very abnormal laboratory test results.
* Have heart, liver, kidney or nervous system conditions.
* Have serious problems digesting and absorbing food or have serious long-term diarrhea within 4
* weeks of randomization.
* Have received radiation (localized is allowed) or chemotherapy within 30 days before randomization.
* Have seizure disorders that cannot be controlled.
* Have received any other drugs that affect the immune system or experimental drugs within 60 days before randomization.
* Have had any vaccination within 15 days before randomization.
* Have a mental condition which makes the patient unable to understand what the study is about and what it involves.
* Have a history of alcohol or drug abuse, unless the investigator feels that it will not interfere with participation in the protocol.
* Are pregnant or breast-feeding.
* Have a history of being very sensitive to the study drug or similar drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - UCSF - San Francisco Gen Hosp, San Francisco, California
  - Northwestern Univ Med School, Chicago, Illinois
  - Univ TX Med Branch, Galveston, Texas